CLINICAL TRIAL: NCT02853279
Title: The Effect of (i) Physical Activity and (ii) Continuous Versus Intermittent Exercise Training Upon Cardiovascular and Cognitive Function in Obese Women
Brief Title: Physical Activity and Intermittent Exercise Training for Cardiovascular and Cognitive Gain in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Karen Birch, Chief Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIOSCI 10-021
Record Dates: First submitted 2016-07-11; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Cognitive Ability, General; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval exercise training (Experimental): Supervised exercise training undertaking interval exercise twice per week for 30 min each visit over 12 weeks.
  Interventions: Behavioral: Interval exercise training
- Continuous exercise training (Active Comparator): Supervised exercise training undertaking continuous exercise twice per week for 30 min each visit over 12 weeks.
  Interventions: Behavioral: Continuous exercise training (CON)

INTERVENTIONS:
Behavioral: Interval exercise training — Interval exercise sessions (INT) involving work:recovery ratios of 40 s at 70% delta work-rate followed by 80 s active recovery at 20 W. 70% delta (∆) is 70% of the difference between work rate peak (WRpeak) and work rate at the lactate threshold (WRLT) calculated as:
  70%∆ =0.7(〖WR〗_peak- 〖WR〗_LT )+ 〖WR〗_LT
  Where WR is work rate, LT is lactate threshold)
  Each session was for 30 min and this was undertaken twice per week for 12 weeks. One home based exercise session was incorporated per week.
  Arms: Interval exercise training
Behavioral: Continuous exercise training (CON) — Exercise sessions involved cycling at 20%∆ work-rate peak for the duration of the session. This work-rate was chosen so that all participants in the group would be exercising in the heavy-intensity domain. To enable participants in the CON exercise group to complete the same amount of work (kJ) as the participants in the INT exercise group, the amount of work that would be completed if the CON participants completed an INT exercise session was calculated. Participants exercised for 26 min (varying to match interval group) twice per week for 12 weeks.
  Arms: Continuous exercise training

SUMMARY:
One hundred participants from a combination of (a) local advertisements and/or (b) those whose details are held on a research database (of previous volunteers indicating willingness to be contacted about future studies) will be sought to volunteer for this study. Written informed consent will be gained following greater than 48 hours for the purpose of reading the Participant Information sheets. The study will then involve two stages (i) recruiting participants for a cross sectional analysis of the relationship between physical activity levels and cardiovascular and cognitive function, and (ii) a longer exercise training study in a subsample of these volunteers (i.e. participants who volunteer to exercise train). Participants for stage 1 will then visit the laboratory in the University on three occasions (over a three week period) to be assessed for body composition, exercise tolerance, current physical activity levels, cognitive function and arterial and cardiac health. Each visit will last for 60 - 90 minutes. Participants will then be provided with an accelerometer to wear for a period of one week in order to assess movement counts and sedentary behaviour. Stage 2 will include only those participants who have volunteered for the exercise training component (approx 60). These participants will then be randomly divided into two groups. Both groups will exercise three times per week for 12 weeks duration. Group 1 will exercise in a traditional manner at a moderate intensity, whilst the second group will exercise at a heavy intensity but in short bursts. Both groups will complete the same amount of work but in two differing modes. Both groups will attend the laboratory twice per week for supervised exercise sessions and also perform one home based 30 minute brisk walk per week. All participants will be re-examined at 12 weeks.

DETAILED DESCRIPTION:
The study will involve two stages (i) recruiting participants for a cross sectional analysis of the relationship between physical activity levels and cardiovascular and cognitive function, and (ii) a longer exercise training study in a subsample of these volunteers. 100 participants for stage 1 will visit the laboratory in the University on three occasions (within a three week period) to be assessed for anthropometric outcomes, body composition, exercise tolerance, cognitive function and arterial and cardiac health. Each visit will last for 60 - 90 minutes. Participants will then be provided with an accelerometer to wear for a period of one week in order to assess movement counts and sedentary behaviour. Stage 2 will include only those participants who are happy to continue into the exercise training phase. These participants will then be matched for age and BMI and then randomly (on matched pairs) allocated to one of two groups. Both groups will exercise three times per week for 12 weeks duration. Group 1 will exercise in a traditional manner undertaking continuous exercise, whilst the Group 2 will exercise at a heavy intensity but in short bursts (interval exercise). Both groups will complete the same amount of work but in two differing modes. Both groups will attend the laboratory twice per week for supervised exercise sessions and also perform one home based 30 minute brisk walk per week. All participants will be re-examined at 12 weeks.

Recruitment of participants

One hundred participants from a combination of (a) local advertisements and/or (b) those whose details are held on a research database (of previous volunteers indicating willingness to be contacted about future studies) will be sought to volunteer for this study. Participants will be contacted via email/telephone/letter to provide information regarding this study. All volunteers interested in participating will be contacted to provide general information during a preliminary telephone screening interview. This will be used to check main inclusion and exclusion criteria. The women who fit these criteria will be sent the participant information sheet to read carefully and if still interested invited to attend the first laboratory visit for a screening session. Participants have greater than 48 hours to assess the participant information sheet before they attend this first visit when, if eligible, they will be asked to provide written informed consent.

Laboratory Visits

Visit 1

During this visit the study and all procedures will be explained in detail to all participants, and written informed consent will be taken. A thorough medical history will be obtained and participants will be asked to complete a Recruitment Information Questionnaire (RIQ) to confirm all inclusion/ exclusion criteria. Participants will complete the National Adult Reading Test (NART) which estimates premorbid intelligence levels.

Participants will also complete a Physical Activity Readiness Questionnaire (PAR-Q) which will be reviewed to determine whether participants are fit to continue with the study. Simple measures of body weight, height and waist circumference will be taken. Participants will complete a practice version of the cognitive test battery to demonstrate the tests, ensure participants understand how to perform the tests correctly and assess compliance (effort).

Participants will complete a cycling test on a stationary bicycle under the supervision of the investigator and a medic.

Visit 2

The second visit will involve several measures of arterial health which requires participants to attend in a 12 hour fasted state. Blood vessel function will be assessed using a blood pressure cuff around the lower arm for a period of 5 minutes. Cardiac structure and function will be assessed using two-dimensional (2D) echocardiography. Vascular function will be assessed using ultrasound and applanation tonometry. All procedures are non-invasive. Percentages of body fat and muscle mass will be measured using bioimpedance.

A 60ml blood sample will be taken which will be used to asses endothelial progenitor cell number and function, insulin sensitivity, cholesterol levels and is part of the assessment for health of the arteries and vascular system.

Visit 3

On the third visit a cognitive function test will be completed, which requires participants to attend in a 12 hour fasted state.

Participants will perform a 45 minute battery of cognitive tests. Following the cognitive tests, participants will be asked to complete a cognitive test evaluation questionnaire to assess both subjective and objective cognition.

At the end of the third laboratory visit all participants will be provided with an ActiHeart accelerometer (Actigraph, Pensacola, USA) to wear for a period of one week in order to assess movement counts and sedentary behaviour. At the end of the seven days the accelerometer is given back to or collected by the team and the data downloaded.

The three baseline laboratory visits plus the seven days using the ActiHeart accelerometer all come under stage 1 of the study. Participants will be asked to continue into the exercise training stage (stage 2), and willing volunteers will move through to the second stage of the experiment. All measures will be repeated at 12 weeks (78 hours to 5 days following cessation of the last exercise training session).

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women (exercise ≤2 day per week)
* Pre-menopausal (age 35- 50 years)
* BMI of ≥30 kg/m2
* Able to give informed consent .
* Non-smokers
* Vision sufficiently good to complete the cognitive testing (using glasses and/or lenses).

Exclusion Criteria:

* Male
* BMI < 30 kg/m2
* Clinically diagnosed with type 1 or type 2 diabetes
* Resting/exercise ECG indicating significant ischemia, recent myocardial infarction or other acute cardiac event or other exercise related ECG abnormalities.
* Unstable angina.
* Uncontrolled hypertension.
* Uncontrolled cardiac dysrhythmias
* The use of antidepressant, antianxiety, or thyroid medication.
* Dementia
* Neurological disorder
* Previous stroke or Transient Ischaemic Attack (TIA)
* Musculoskeletal impairment or injury
* Medication that has a direct effect on the brain and is likely to influence cognitive function.
* Current smokers or those who have given up in the previous 6 months

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake (CPX) | Change at 12 weeks
  Maximal oxygen uptake assessed during a ramp incremental cycle ergometry test.
Flow mediated dilatation | Change at 12 weeks
  Percentage change in brachial artery diameter following cuff occlusion using doppler ultrasound.

SECONDARY OUTCOMES:
Lactate threshold | Baseline and 12 weeks
  Lactate threshold estimated from pulmonary gas exchange criteria
Blood borne (plasma) inflammatory marker | Baseline and 12 weeks
  high sensitivity C reactive protein
Work rate peak | Baseline and 12 weeks
  The peak work rate achieved during the maximal oxygen uptake assessment
Circulating angiogenic cell number | Baseline and 12 weeks
  CD34+CD45dimKDR+ via Flow cytometry
Circulating cytokines | Baseline and 12 weeks
  vascular endothelial growth factor
Circulating cytokines | Baseline and 12 weeks
  stromal derived factor 1
Arterial stiffness | Baseline and 12 weeks
  Doppler assessed and Sphygmacor assessed changes in stiffness via pulse wave velocity
Cognitive function (Visual spatial learning scale) | Baseline and 12 weeks
Cognitive function (Tower of Hanoi) | Baseline and 12 weeks
Cognitive function (Grooved peg board) | Baseline and 12 weeks
Cognitive function (Visual verbal learning scale) | Baseline and 12 weeks
Cognitive function (Bakan test)) | Baseline and 12 weeks
Cognitive function (Corsi block tapping) | Baseline and 12 weeks
Physical activity level | Baseline and 12 weeks
  Accelerometer assessed physical activity (Actiheart) worn on the hip
Blood pressure | Baseline and 12 weeks
  Blood pressure
Body composition | Baseline and 12 weeks
  Bioelectrical impedence analysis (BIOSTAT) assessment of fat mass
Cardiac function (echocardiography) | Baseline and 12 weeks
Cardiac structure (echocardiography) | Baseline and 12 weeks
Adhesion of cultured angiogenic cells to vascular smooth muscle cells | Baseline and 12 weeks
  Number of cells adhering

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Birch, PhD, Principal Investigator — University of Leeds
Locations (2):
- United Kingdom (2):
  - Centre for Sports and Exercise Sciences, University of Leeds, Leeds, West Yorkshire
  - Human Appetite Research Unit, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 3 abstracts presented to the annual congress of the European College of Sports and Exercise Sciences, Barcelona, Spain, 2013 — http://www.vlgafc.ru/files/s/1ECSSBABS2013.pdf